CLINICAL TRIAL: NCT00861848
Title: Quantification of Ventricular Mechanics/Myocardial Blood Flow Reserve in Adolescents and Adults Ages 12-50 With Congenital or Acquired Heart Disease Using Bicycle Stress With Real Time Myocardial Contrast Echo and Dobutamine Stress MRI
Brief Title: Real Time Myocardial Contrast Echocardiography and Dobutamine Stress Perfusion Magnetic Resonance Imaging
Acronym: ECHOBIKE
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0599-08-FB
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Kawasaki Disease; Heart Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 12-50 with heart disease: 12-50 with heart disease
- 12-50 normal controls: 12-50 normal controls

SUMMARY:
The present study is designed to:

1. investigate the safety and efficacy of Real time myocardial echocardiography (RT-MCE) in adolescents and adults ages 12-50 with congenital and acquired congenital heart disease
2. compare RT-MCE with dobutamine stress perfusion MR for determination of coronary flow reserve and ventricular wall motion
3. assess regional myocardial mechanics using myocardial speckle tracking and MR tagging.
4. evaluate RV volume and function for a subset of subjects using novel reconstruction software

DETAILED DESCRIPTION:
Individuals will be identified from the cardiology database and consented during their routine follow up visits. Exercise stress, transthoracic echocardiography and cardiac MR are part of standard medical care in the follow up evaluation of adolescents and adults with repaired congenital heart disease. The use of contrast (with transthoracic echocardiography) and dobutamine stress testing (with the cardiac MR) will be performed as part of the research study. After signing consent/ assent, a study subject will have pertinent medical history (e.g. past palliation and operative repair dates and type, current medications, review of systems) and physical exam findings extracted from the medical record, especially the recording of the most recent clinic visit. If the subject is a female of child bearing age, a serum pregnancy test will be done at this time. This data will be recorded using standardized case report forms for history and physical exam. The study patients will complete a standardized interview to determine their exercise tolerance according to New York Heart Association (NYHA) classification. All patients who consent to the additional testing will require an additional 1 hour of time to the regular Echo and CMR testing.

Each patient will have the protocol supine bicycle stress with contrast echocardiogram performed at UNMC Echo lab.. The study subject will then have the clinically indicated CMR study (Philips Achieva 1.5T magnet), scheduled and performed by a qualified CMR technologist, working with a pediatric or adult cardiologist. An attempt will be made to have CMR and Echo performed on the same day to minimize physiologic variability, but will at least be done within 1 week each other. Further post-processing (wall motion analyses, speckle tracking and myocardial tagging) and image analyses will be performed by the principal investigators on standard workstations.

ELIGIBILITY:
Inclusion Criteria:• Age between 12 years and 50 years.

* Male or female.
* History of repaired congenital heart disease including atrial septal defects, aortic valve disease, tetralogy of fallot, transposition of great arteries and anomalous left coronary artery from pulmonary artery.
* History of sequelae of heart disease acquired as an infant or child, including Kawasaki disease and coronary ectasia, and patients post anthracycline chemotherapy.
* Ability to perform Supine bicycle stress with contrast echocardiography as determined by primary cardiologist and/or Dr. Shelby Kutty.
* Ability to perform CMR with dobutamine stress as determined by the patients primary cardiologist and/or Dr. Shelby Kutty
* Signed informed consent and assent as applicable.

Exclusion Criteria:• Atrial or ventricular arrythmias that cannot be controlled to heart rates < 70/min

* Intracardiac shunts
* Known hypersensitivity to perflutren
* Known hypersensitivity to Dobutamine
* Congestive heart failure in NYHA class II, III or IV
* Claustrophobia or any other reason patient is unable to perform CMR (i.e. ferromagnetic implants causing significant artifact that alters image quality, presence of pacemaker, AICD, etc.)
* Pregnant or possibly pregnant (based on history/information obtained from the patient) or breast feeding

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: ages 12-50 with congenital and acquired congenital heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
The present study is designed to: (1) investigate the safety and efficacy of Real time myocardial echocardiography (RT-MCE) in adolescents and adults ages 13-40 with congenital and acquired congenital heart disease. | 2 years
  The present study is designed to: (1) investigate the safety and efficacy of Real time myocardial echocardiography (RT-MCE) in adolescents and adults ages 13-40 with congenital and acquired congenital heart disease.

SECONDARY OUTCOMES:
Compare RT-MCE with dobutamine stress perfusion MR for determination of coronary flow reserve and ventricular wall motion (3) assess regional myocardial mechanics using myocardial speckle tracking and MR tagging. | 2 years
  Compare RT-MCE with dobutamine stress perfusion MR for determination of coronary flow reserve and ventricular wall motion (3) assess regional myocardial mechanics using myocardial speckle tracking and MR tagging.

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Kutty, MD, Principal Investigator — UNMC; Thomas Porter, MD, Principal Investigator — UNMC
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kutty S, Olson J, Danford CJ, Sandene EK, Xie F, Fletcher SE, Erickson CC, Kugler JD, Danford DA, Porter TR. Ultrasound contrast and real-time perfusion in conjunction with supine bicycle stress echocardiography for comprehensive evaluation of surgically corrected congenital heart disease. Eur Heart J Cardiovasc Imaging. 2012 Jun;13(6):500-9. doi: 10.1093/ejechocard/jer287. Epub 2011 Dec 15. PMID 22173935